CLINICAL TRIAL: NCT02527213
Title: Randomized Double Blind Placebo Controlled Trial of Sodium Thiosulfate for the Treatment of Pain Associated With Calcific Uremic Arteriolopathy Followed by a Single Armed Extension Phase to Prospectively Observe Lesion Progression
Brief Title: Double-blind Trial of Sodium Thiosulfate for the Treatment of Pain Associated With Calcific Uremic Arteriolopathy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision -terminated on 30 October 2015
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1STS12001
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Calciphylaxis; Calcific Uremic Arteriolopathy
MeSH Terms: conditions — Calciphylaxis | interventions — sodium thiosulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Thiosulfate (Experimental): Sodium Thiosulfate at 25g in 100 ml normal sterile saline (NSS)
  Interventions: Drug: Sodium thiosulfate
- Placebo (Placebo Comparator): similarly-formulated placebo in 100 ml NSS
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium thiosulfate — Additional treatment(s) due to lesion progression When intervention occurs, the date of the intervening event should be recorded in the source documents and the (CRF). The subject should continue in the study as scheduled.
  Arms: Sodium Thiosulfate
Drug: Placebo — Additional treatment(s) due to lesion progression When intervention occurs, the date of the intervening event should be recorded in the source documents and the (CRF). The subject should continue in the study as scheduled.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of Sodium Thiosulfate (STS) compared to placebo, in reducing analgesic requirement in subjects with calcific uremic arteriolopathy (CUA) during an initial 28-day treatment phase.

DETAILED DESCRIPTION:
Efficacy of Sodium Thiosulfate (STS) compared to placebo, in reducing analgesic requirement in subjects with calcific uremic arteriolopathy (CUA) during an initial 28-day treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age who are able to give informed consent.
2. Calcific uremic arteriolopathy (CUA), either newly-diagnosed or pre-existing, currently on STS or not yet treated with STS and either not on pain medication or on a stable pain medication regimen. The diagnosis of calciphylaxis can be made when:

   * The following clinical features are all present, or two (2) of the following clinical features and typical histopathological findings are present.

Clinical features:

1. A patient on chronic hemodialysis for chronic kidney disease or with a glomerular filtration rate (GFR) of less than 15/ml/min/1.73 m2
2. More than 2 painful and non-treatable skin ulcers with concomitant painful purpura
3. Painful and non-treatable skin ulcers on the trunk, extremities, or penis with concomitant painful purpura

Histopathological findings by skin biopsy when 3 clinical findings are not present:

1. Necrosis and ulceration of the skin with calcification of the tunica media and internal elastic membrane of small to medium-sized arterioles of dermis and subcutaneous fat are essential for the diagnosis
2. Concentric stenosis due to edematous intimal thickening is also seen in the small to medium-sized arterioles of dermis and subcutaneous fat
3. End stage renal disease (ESRD) on chronic maintenance hemodialysis.
4. Willingness to undergo washout of pre-existing STS treatment (if required by treatment allocation) and to continue in a double blind treatment period of 4 weeks, during which they might receive placebo.
5. Ability to comply with all study requirements.

Exclusion Criteria:

1. History of allergic or other adverse reaction to STS
2. Current treatment with STS for indications other than CUA (e.g. cyanide poisoning)
3. Currently on alternative treatment for CUA as listed below. Unless treatment has been discontinued for at least 1 month prior to the screening visit.

   1. Steroids
   2. Hyperbaric Oxygen
   3. Bisphosphonates
   4. Pentoxifylline
   5. Tissue Plasminogen Activator
   6. Lucilia sericata larvae (maggot therapy)
   7. On Cinacalcet for treatment for CUA (i.e. cinacalcet was either started or dose increased after the appearance of lesions)
4. Any co-existing disease or problem that makes participation in the study unadvisable for the patient or compromises integrity of the study

   1. Cirrhosis of the liver
   2. History of congestive heart failure (New York Heart Association class III or IV) with multiple hospital admissions (at least 3 admissions in 6 months)
   3. Persistent and uncontrolled metabolic acidosis
5. Chronic kidney disease or renal transplant patients with diagnosis of calciphylaxis who are not on hemodialysis.
6. Any other disease or condition which, in the judgment of the Investigator, would place a subject at undue risk by being enrolled in the trial, or cause inability to comply with the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-30 (Estimated); Primary Completion 2016-08-29 (Estimated); Study Completion 2016-08-29 (Estimated)

PRIMARY OUTCOMES:
Reduction in Analgesic Requirement | up to 28 Days
  The length of time in days, from first treatment with blinded study drug; to when subject requires rescue analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mundy, MD, PhD, Study Director — American Regent, Inc.
Locations (3):
- United States (3):
  - Nephrology Consultants, Huntsville, Alabama
  - Nephrology Association of Northern Indiana, Fort Wayne, Indiana
  - A.A. Northeast Clinical Research Center, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No